CLINICAL TRIAL: NCT00659126
Title: A Phase II Study of Ferumoxytol and Gadolinium Magnetic Resonance Imaging at 3T and 7T in Subjects With Primary or Metastatic Brain Tumors Either Before or After Therapy
Brief Title: Ferumoxytol- and Gadolinium-Labeled MRI in Measuring Tumors Before or After Treatment in Patients With Primary or Metastatic Brain Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Edward Neuwelt, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00002864; NCI-2015-00225 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SOL-06077-L; IRB00002864 (Other: OHSU Knight Cancer Institute); R01CA137488 (NIH)
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Malignant Neoplasm in the Brain; Primary Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Ferrosoferric Oxide; Gadolinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (Gd, ferumoxytol, 3T or 7T MRI) (Experimental): Patients receive gadolinium IV on day 1 and ferumoxytol non-stoichiometric magnetite IV on day 2. Patients undergo anatomical MRI sequences with 3T or 7T at baseline and on days 1-3. Patients also undergo DSC MRI and DCE MRI on days 1-2. Day 1 and day 2 imaging sessions may be separated by up to 7 days.
  Interventions: Procedure: 3 Tesla Magnetic Resonance Imaging; Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Procedure: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging; Drug: Ferumoxytol; Drug: Gadolinium; Procedure: High Field Strength Magnetic Resonance Imaging; Procedure: Susceptibility Weighted Imaging

INTERVENTIONS:
Procedure: 3 Tesla Magnetic Resonance Imaging — Undergo 3T MRI
  Other Names: 3 Tesla MRI; 3T MRI
Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging — Undergo DCE MRI
  Other Names: DCE MRI; DCE-MRI; DYNAMIC CONTRAST ENHANCED MRI
Procedure: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging — Undergo DSC MRI
  Other Names: DSC-MRI; Dynamic Susceptibility Contrast-Enhanced MRI; DYNAMIC SUSCEPTIBILITY-CONTRAST MRI
Drug: Ferumoxytol — Given IV
  Other Names: Feraheme; Ferumoxytol Non-Stoichiometric Magnetite
Drug: Gadolinium — Given IV
  Other Names: Gd
Procedure: High Field Strength Magnetic Resonance Imaging — Undergo 7T MRI
  Other Names: High Field Strength MRI
Procedure: Susceptibility Weighted Imaging — Undergo SWI
  Other Names: BOLD Venographic Imaging; BOLD Venography; SWI

SUMMARY:
This phase II trial studies how well magnetic resonance imaging (MRI) using contrast imaging agent ferumoxytol works in comparison to standard imaging agent gadolinium in measuring tumors in patients undergoing treatment for brain tumors or other tumors that have spread to the brain. Diagnostic procedures, such as MRI, may help find and diagnose disease and find out how far the disease has spread. MRI scans use radio waves and a powerful magnet linked to a computer to create detailed pictures of areas inside the body. The contrast imaging agent ferumoxytol consists of small iron particles taken by the blood stream to the brain and to the area of the tumor. It is highly visible on the MRI, and may help visualize the blood flow going through the tumor better than gadolinium can. Using a more sensitive and faster 7 Tesla (7T) magnet MRI in conjunction with a contrast imaging agent may provide a better way to measure tumors than the 3 Tesla (3T) magnet MRI in patients with brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare quantitative blood brain barrier permeability measurements (derived transfer coefficient [Ktrans]) of a standard gadolinium (Gd) MRI contrast agent at 3T and 7T using dynamic contrast enhancement (DCE) MRI.

II. To compare dynamic susceptibility contrast (DSC) based perfusion measures at 3T and 7T.

SECONDARY OBJECTIVES:

I. To describe the blood brain barrier permeability to ferumoxytol (ferumoxytol non-stoichiometric magnetite) and to a standard gadolinium-based MRI contrast agent using signal intensity changes as described above.

II. To describe cerebral blood volume (CBV) measurements obtained using a standard gadolinium MRI contrast agent and ferumoxytol.

III. To evaluate tumor microvascularity on susceptibility-weighted images (SWI).

IV. To describe the microscopic distribution of ferumoxytol particles in tissue removed from subjects undergoing surgery.

OUTLINE: Patients are assigned to 3T or 7T magnet within the subgroups.

Patients receive gadolinium intravenously (IV) on day 1 and ferumoxytol non-stoichiometric magnetite IV on day 2. Patients undergo anatomical MRI sequences with 3T or 7T at baseline and on days 1-3. Patients also undergo DSC MRI and DCE MRI on days 1-2. Day 1 and day 2 imaging sessions may be separated by up to 7 days.

After completion of study, patients are followed up at approximately 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with radiographically suspected, histologically or cytologically confirmed primary brain tumors or brain metastasis are eligible
* Subjects may be enrolled at any point in diagnosis or treatment
* Subjects must have had radiographically evaluable or measurable disease with standard magnetic resonance (MR) imaging
* Members of all races and ethnic groups will be included
* Eastern Cooperative Oncology Group (ECOG) performance status =< 3 (Karnofsky performance status [KPS] >= 30)
* Ability to understand and the willingness to sign a written informed consent document, or have a representative able to consent for the subject
* Sexually active women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study treatment and for the duration of study treatment; should a female become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Subject agrees to complete follow up visit

Exclusion Criteria:

* Subjects with clinically significant signs of uncal herniation, such as acute pupillary enlargement, rapidly developing motor changes (over hours), or rapidly decreasing level of consciousness
* Subjects who have a contraindication for MRI: metal in their bodies (a cardiac pacemaker or other incompatible device), are severely agitated, need monitored anesthesia for scanning, or have an allergy to Gd contrast material
* Subjects with known hepatic insufficiency or cirrhosis
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ferumoxytol
* Subjects with known or suspected iron overload (genetic hemochromatosis or history of multiple transfusions)
* Subjects expecting to undergo surgery between the imaging sessions; subjects may undergo surgery at any time before the first, or after the last imaging session; this exclusion only applies to each study visit (3 day scanning session), and does not apply to the time (at least 3 weeks) between each study visit
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating women are excluded from this study
* Inability or unwillingness to undergo the complete series of imaging sessions; inability or unwillingness to complete the one month follow-up
* Human immunodeficiency virus (HIV)-positive subjects on combination antiretroviral therapy are ineligible
* Subjects with glomerular filtration rate (GFR) < 50
* Subjects with three or more drug allergies from separate drug classes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-11-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Neuwelt, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 3 Tesla in Subjects With Brain Tumors: A subset of subjects with primary or metastatic brain tumors will be assigned to 3 Tesla MRI and will undergo gadolinium enhanced imaging on day 1, ferumoxytol enhanced imaging on day 2, and a non contrast ("post-ferumoxytol") imaging on day 3. All scans will be performed on a 3 Tesla MRI scanner.
- Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 7 Tesla in Subjects With Brain Tumors: A subset of subjects with primary or metastatic brain tumors will be assigned to 7 Tesla MRI and will undergo gadolinium enhanced imaging on day 1, ferumoxytol enhanced imaging on day 2, and a non contrast ("post-ferumoxytol") imaging on day 3. All scans will be performed on a 7 Tesla MRI scanner.
Period: Overall Study
Arm/Group | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 3 Tesla in Subjects With Brain Tumors | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 7 Tesla in Subjects With Brain Tumors
Started | 15 | 25
Completed | 12 | 21
Not Completed | 3 | 4
Not completed — Adverse Event | 2 | 2
Not completed — Screen failure | 1 | 1
Not completed — Technical problems with MRI | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 3 Tesla in Subjects With Brain Tumors | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 7 Tesla in Subjects With Brain Tumors | Total
Number analyzed (Participants) | 15 | 25 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (12.91) | 52.52 (13.69) | 53.45 (13.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 14
  Male | 11 | 15 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 13 | 24 | 37
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 25 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Brain tumor type [Count of Participants; unit: Participants]
  Glioblastoma | 8 | 8 | 16
  Anaplastic astrocytoma | 2 | 5 | 7
  Astrocytoma grade II | 1 | 0 | 1
  Anaplastic oligodendroglioma | 0 | 1 | 1
  Oligodendroglioma grade II | 0 | 4 | 4
  Meningioma | 1 | 3 | 4
  Metastasis | 0 | 0 | 0
  CNS lymphoma | 1 | 0 | 1
  Other | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Contrast to Noise Ratio (CNR), in Terms of Normalized Signal Intensity Changes, for T1-weighted MRI Signal at 3T and 7T (Gadolinium [Gd] T1-weighted Magnetic Resonance Imaging [MRI] DCE Data Only)
Description: Paired sample t-tests will be used for primary descriptive comparisons. Secondary analyses will use a repeated measures analysis of variance (ANOVA) model to compare 3T and 7T while adjusting for other factors including tumor type, prior therapy, and, potentially, important baseline factors that differ between the subjects assigned to the two field strengths. Normality will be assessed graphically and, if needed, a transformation (e.g. the logarithmic transform) will be applied.
Time Frame: Baseline to day 1
Population: The first primary objective was to use dynamic contrast enhancement (DCE) MRI. Due to limitations of the scanners, these images were not collected. Dynamic susceptibility contrast (DSC) images were collected which are reported in the second primary objective.
Arm/Group | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 3 Tesla in Subjects With Brain Tumors | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 7 Tesla in Subjects With Brain Tumors
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: CNR, in Terms of Normalized Signal Intensity Changes, for Dynamic Susceptibility Contrast (DSC) MRI Data Sets at 3T and 7T (Gadolinium and Ferumoxytol)
Description: A two sample t-test was used for primary descriptive comparisons since CNR was measured on different subjects at 3T and 7T. There were no repeated measures in the resulting data. Given the small sample size, a linear regression was conducted to compare CNR between 3T and 7T only adjusted for Fe dose. No other adjusted analyses were conducted.
  CNR was compared between 3T and 7T for both Ferumoxytol and Gadolinum. Ferumoxytol was administered using three injections and CNR was measured after each injection, thus we have three measures of CNR (Fe1CNR, Fe2CNR and Fe3CNR).
Time Frame: Day 1 to day 2
Population: Other patients were excluded due to poor DSC graph or no residual tumor for measurement or residual tumor stayed within vascular lumen. Non-contrast (day 3) data not collected.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 3 Tesla in Subjects With Brain Tumors | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 7 Tesla in Subjects With Brain Tumors
Number analyzed (Participants) | 10 | 10
ratio
  Gadolinium | 1.34 (.923) | .912 (.519)
  Ferumoxytol 1st dose | 1.034 (.611) | .669 (.644)
  Ferumoxytol 2nd dose | 1.27 (.886) | 1.08 (1.15)
  Ferumoxytol 3rd dose | 1.45 (.893) | .886 (.964)

3. Secondary Outcome: Relevant Dynamic MRI (Dynamic Contrast Enhancement [DCE] and DSC) Signal Intensity Changes for Permeability and Perfusion
Description: Mixed model repeated measures ANOVAs will be fit. Factors will include imaging agent (Gd or ferumoxytol) and field strength (3T and 7T). Each subject will contribute one measure for each combination of imaging agent and field strength (4 measures total).
Time Frame: Day 1 to day 2
Population: Data for secondary outcomes were not collected. The study was terminated early as the 7t scanner was not providing the images needed, and we did not have the funding to continue.
Arm/Group | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 3 Tesla in Subjects With Brain Tumors | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 7 Tesla in Subjects With Brain Tumors
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Cerebral Blood Volume (CBV) Measurements, Quantified Using DSC Techniques
Description: Blood volumes will be compared using repeated measures ANOVA to compare the imaging agents.
Time Frame: Day 1 to day 2
Population: as for outcome 3
Arm/Group | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 3 Tesla in Subjects With Brain Tumors | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 7 Tesla in Subjects With Brain Tumors
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Tumor Microvascularity on Susceptibility-weighted Images (SWI) Before and After Ferumoxytol
Description: Analysis will also include covariates of prior therapy. For the comparisons between treated and untreated subjects, means and confidence intervals will be estimated for each group for the perfusion and permeability measures and for the baseline characteristics.
Time Frame: Day 1 to day 2
Population: as for outcome 3
Arm/Group | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 3 Tesla in Subjects With Brain Tumors | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 7 Tesla in Subjects With Brain Tumors
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Presence of Iron Staining
Description: The pathology will be analyzed qualitatively for the presence of iron staining. The amount and localization of the staining will be assessed, with attention paid to whether the tumor cells themselves or reactive cells in and around the tumor demonstrate iron uptake.
Time Frame: At time of surgery
Population: as for outcome 3
Arm/Group | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 3 Tesla in Subjects With Brain Tumors | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 7 Tesla in Subjects With Brain Tumors
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events from day 1 of imaging session to 4 to 6 weeks after completing imaging.
Description: Non-contrast (day 3) data not collected.
Arm/Group | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 3 Tesla in Subjects With Brain Tumors | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 7 Tesla in Subjects With Brain Tumors
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/21
Other Adverse Events (participants affected / at risk) | 0/12 | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 3 Tesla in Subjects With Brain Tumors (N=12) | Gadolinium and Ferumoxytol Magnetic Resonance Imaging at 7 Tesla in Subjects With Brain Tumors (N=21)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT00659126/Prot_SAP_ICF_000.pdf